CLINICAL TRIAL: NCT06263465
Title: Precision Vaginal Microbiome Transplantation in Women With Bacterial Vaginosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: ZhuHai Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Zhou, Professor, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CALM
Record Dates: First submitted 2024-01-23; First posted 2024-02-16 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus cispatus (Experimental): 10^9 cfu,5 days
  Interventions: Other: Lactobacillus cispatus
- Placebo (Placebo Comparator): 0 cfu,5 days
  Interventions: Other: placebo

INTERVENTIONS:
Other: Lactobacillus cispatus — 10^9 cfu,5 days
  Arms: Lactobacillus cispatus
Other: placebo — 0 cfu,5 days
  Arms: Placebo

SUMMARY:
The aim of this study was to explore the efficacy and safety of a new vaginal microbiome transplantation technique, using Lactobacillus cispatus from healthy donors as a treatment of bacterial vaginosis.

DETAILED DESCRIPTION:
The volunteers will be recruited from the women who come to the hospital to do the bacterial vaginosis test. After being informed about the potential risks, each volunteer giving written informed consent will be asked to complete a questionnaire.

Then, posterior fornix of vagina secretions will be taken from each volunteer to perform 16S rRNA gene sequencing microecology assessment , Clue cell detection and amine test.

After 2weeks ,1 month ,3 months,6 months,12 monthssince the entry, each volunteer will be asked to go back to research center to do the same sampling and examination as previously did in entry.

ELIGIBILITY:
Inclusion Criteria:

1. History of sexual behaviour 2.18-55 years old 3. Women were diagnosed as bacterial vaginosis

Exclusion Criteria:

1. During pregnancy, or within 8 weeks after delivery;
2. presence of systemic diseases (such as SLE, malignant tumors, etc.)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BV recurrence rate | month 12
  Primary Outcome Measure

SECONDARY OUTCOMES:
vaginal secretions 16s rRNA gene sequencing | 2 weeks，month 1，month 3、month 6、month 12
  Secondary Outcome Measures
BV recurrence rate | 2 weeks，month 1，month 3、month 6
  Secondary Outcome Measures

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Principal Investigator — Department of Laboratory Medicine, Zhujiang Hospital, Southern Medical University
Locations (1):
- Zhuhai People'S Hospital, Zhuhai, Guangdong, China